CLINICAL TRIAL: NCT00333879
Title: Virtual Reality Mobility Training System for Veterans With Vision Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: C4188-R
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Blindness
Keywords: Rehabilitation; Sensory Aid
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual Sound System (Other): Efficacy of using a virtual sound system to simulate street crossing conditions.
  Interventions: Device: Virtual Sound System

INTERVENTIONS:
Device: Virtual Sound System — Virtual Sound System is tested for efficacy in its ability to realistically simulate Street Crossings sounds in a safe indoor environment. If efficacious, Blind students will be able to practice crossing streets in safety indoors.
  Other Names: 3-D Sound Simulation System

SUMMARY:
This is a two-year proof-of-concept study to evaluate a new Virtual Reality (VR) "holographic" sound system for use as an audiological Orientation and Mobility (O&M) training tool

DETAILED DESCRIPTION:
This is a two-year proof-of-concept study to evaluate a new Virtual Reality (VR) "holographic" sound system for use as an audiological Orientation and Mobility (O&M) training tool. This new system avoids the limitations of other technologies (i.e., binaural recordings and existing VR sound systems) that have been employed with limited success for audiological training. Four advancements in the state-of-the-art represented by this new holographic system provide new promise for audiological O&M training. First, unlike binaural systems, the new system allows the person to move their head in a natural fashion to localize sounds. Second, a spherical microphone array is used to record sound environments so as to retain the direction from which each ambient sound originated. When these recorded sound environments are later presented through head-tracking headphones in a VR environment, real-time software maintains the directionality of the sound so that it remains true no matter how the person moves or turns their head. Third, this new system models the actual physical acoustic structure of each person's head and ears to present sounds as they would be heard by that particular person in the recorded setting. Fourth, this system uses software algorithms to isolate specific sounds (i.e., of a moving vehicle) so that during virtual playback, these sounds can be inserted into the virtual sound field at will and in a customizable fashion to create truly unique and flexible virtual sound presentations.

There are two study hypotheses. First, when using sounds to negotiate traffic intersections, skills employed by experienced travelers in real environments will readily transfer to the proposed VR environment to the extent that audiological tasks performed in real environments are just as easily performed in the VR environment. Second, when the VR environment is enhanced to emphasize critical sound cues and eliminate distracting or confusing noises and sounds, performance by skilled travelers in the VR environment will be significantly better than in the actual environment.

The objectives are to: (1) adapt the existing spherical microphone array and digital recording software algorithms to best suit the capture of critical intersection sounds used for intersection negotiations; (2) develop software algorithms to deconstruct intersection sounds, isolating each sound for the VR construction of specific environments of varying complexity; (3) determine the level of sound detail necessary for negotiating intersections successfully; (4) expand the existing system to obtain the desired level of detail; (5) develop software to provide the ability to control the relative emphasis of a variety of sound elements being presented so as to simplify the auditory task; and (6) employ study participants to compare performance in the VR environment with outdoor performance.

Once validated, this system should be able to: (1) leverage instructor time by providing students with an effective means of practicing audiological skills on their own, (2) provide instructors with a means of introducing concepts in a graduated learning sequence that is not dependent on the happenstance availability of specific sounds and conditions found in real environments, and (3) provide audiological training for environments not located in the vicinity of the training site, but which do represent the veteran's home community.

Research will be conducted in collaboration with investigators in the Perceptual Interfaces and Reality Laboratory (PIRL) at the University of Maryland who initially conceived and developed this holographic VR sound system.

COMPARISONS: Outdoor O&M training exclusively

ELIGIBILITY:
Inclusion Criteria:

* Must have little or no light perception
* OMCT (Orientation-Memory Concentration Test) of 10 or less
* Must have been independently and regularly crossing busy intersections for at least 3 years
* Ambulatory and able to walk for at least 10 minutes at a time without resting
* Auditory function at 25 db HL

Exclusion Criteria:

* Imbalance between ears - HL difference of 20 db HL or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Ross, MSEE Med, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 4 totally blind Participants were recruited over three months (April - June) 2009 from the Atlanta Center for Visual Impairment.
Pre-assignment Details: All 4 subjects were accepted for the study. None were excluded.
Period: Overall Study
Arm/Group | Virtual Sound System
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Sound System
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Accuracy in Judging Direction of Traffic at Traffic Intersection
Description: Standing at an intersection subject indicates when traffic is moving left to right and right to left in front of him, versus traffic moving to and away on the street parallel to his path. Subject can respond in only two ways: 1) traffic is moving on the street in front of me, or 2) traffic is moving on the street beside me.
  Each trial lasts 5 minutes with a 2 minute and 30 second break between trials. Traffic stops and starts 5 times over the 5 minutes, each time moving in one of two randomly selected directions: 1) left and right in front of the subject, or 2) forward and back along the street beside the subject.
  The participant must correctly state the direction of traffic at least 4 out of five times for the equipment under test to be counted as efficacious for presenting accurate 3D sound information to the participant.
Time Frame: 4 trials over 30 minutes after 30 minutes of training
Population: Initial pilot study design called for 16 subjects to provide data of significance based on a power analysis. Study terminated at 4 subjects when none of the subjects could identify the location of traffic vehicles when using the intervention across multiple (4) trials.
Measure: Number; unit: participants
Arm/Group | Virtual Sound System
Number analyzed (Participants) | 4
participants | 0

2. Secondary Outcome: Accuracy in Selecting Appropriate Time to Cross Street
Description: Subject is able to state when it is safe to cross the street based on traffic on the street beside him accelerating into motion after traffic on the street in front of him coming to a stop. Subject must state is it safe to cross within 5 seconds of the cars on the street beside him accelerating into motion.
  The system under test will be considered efficacious if the subject is correct at least 4 out of 5 times. This counts as being efficacious for that one subject.
Time Frame: 4 trials over 30 minutes after 30 minutes of training
Measure: Number; unit: participants
Arm/Group | Virtual Sound System
Number analyzed (Participants) | 4
participants | 0

ADVERSE EVENTS:
Arm/Group | Virtual Sound System
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Technical problems with Virtual Sound System. None of the first 4 Subjects could distinguish between sounds in front versus sounds beside them.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes